CLINICAL TRIAL: NCT07149844
Title: Comparing the Effects of Tea Tree Oil (Melaleuca Alternifolia) and Conventional Topical Dressing on Healing of Second-Degree Burn Wounds
Brief Title: Healing Effect of Tea Tree Oil on Burn
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1482025
Record Dates: First submitted 2025-08-18; First posted 2025-09-02 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-08

CONDITIONS: Burn
Keywords: Burn; Tea Tree Oil
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- conventional dressing (Other): Conventional dressing: Is the routine study hospital's burn dressing technique, utilizing sterile topical gauze dressing that is impregnated with or laid over a topical antibacterial, silver sulphadiazin dressing secured with adhesive tape.
  Interventions: Drug: tea tree oil ointment

INTERVENTIONS:
Drug: tea tree oil ointment — Petrolatum (petroleum jelly) was sterilized in the oven at 160°C for 90 min, then The ointment was prepared as 10% .
  Other Names: فtea tree ointment

SUMMARY:
Tea tree oil (TTO) has been recognized for its effectiveness in treating infected burns, insect bites, and promoting wound healing. This clinical study aimed to compare the impact of Tea tree oil dressings versus conventional ones in the healing process of second degree burns wounds.

DETAILED DESCRIPTION:
This quasi-experimental comparative controlled clinical trial was conducted at the Burn Unit of Ras-Elteen General Hospital in Alexandria, Egypt. A purposive sample of 30 adult patients with second-degree burns on the chest, abdomen, upper limbs (excluding hands), and lower limbs (excluding feet) was enrolled from the Emergency and Outpatient Departments. Participants were sequentially assigned to two equal groups:

Control group (n=15): Received conventional dressings (sterile gauze with silver sulfadiazine).

Study group (n=15): Received topical 10% tea tree oil (TTO) ointment applied directly to wounds.Wounds were cleansed with sterile normal saline (0.9%), and non-viable tissue was debrided.

Dressings were changed every other day unless soiled or damp. Burns near joints were maintained in functional positions.Wound assessment was performed on days 7, 14, and 21 post-treatment

ELIGIBILITY:
Inclusion Criteria:

* Patient willing to participate and communicate
* Newly admitted with recent 2nd-degree burns (superficial or deep) involving ≤10% of TBSA
* Length of hospital stay of 10 days

Exclusion Criteria:

Any associated illnesses that may affect wound healing, such as:

* Diabetes mellitus (DM)
* Immune disorders
* Pre-existing skin conditions (e.g., eczema)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-07-02 (Actual); Primary Completion 2023-07-22 (Actual); Study Completion 2023-09-22 (Actual)

PRIMARY OUTCOMES:
morphological wound changes | 3 weeks
  assessment of: wound bed, wound margin: color, size, depth, presence of exudates: its amount, color, odor, and type, or scare, edema and granulation tissue formation; in addition to assessment of the wound's surrounding skin condition for: erythema, hotness, tenderness, swelling, separation of deep tissues, fever and peri-wound skin laceration. Each item was rated to score on 2 points Likert scale: 0 = not present and 1= Present.
  A total score of every patient in both groups was summed up and converted into percent score. to desribe wound healing process as ; complete healing: ; Partial healing: and No healing: where higher percent represent better healing
Local infection scoring system | 3 weeks
  Local infection scoring system was recorded as: 0= Absence of infection. 1= Presence of local signs of wound infection (redness, hotness, tenderness, purulent discharge and swelling)2 = Presence of systemic wound infection signs (fever, elevated WBCs, ESR and elevated CRP)

CONTACTS AND LOCATIONS:
Overall Officials: hoda fathy, prof, Principal Investigator — Alexandria University
Locations (1):
- Ras Eltin Hospital, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes
data can be shared on researchgate or other official database
Supporting Information: Study Protocol, SAP
Time Frame: upon acceptance of the manuscript
Access Criteria: upon request

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-10): https://cdn.clinicaltrials.gov/large-docs/44/NCT07149844/Prot_SAP_000.pdf